CLINICAL TRIAL: NCT00228683
Title: Hepatoblastoma Biology Study and Tissue Bank
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: national study, local site not responsible for any analysis/results/etc
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Howard Katzenstein, Associate Professor, Emory University
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: IRB00024899
Record Dates: First submitted 2005-09-27; First posted 2005-09-29 (Estimated); Last update posted 2013-11-26 (Estimated); Status verified 2013-11

CONDITIONS: Hepatoblastoma
MeSH Terms: conditions — Hepatoblastoma | interventions — Tissue Banks

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Biology Study and Tissue Banking — Collection of specimens from Hepatoblastoma patients.

SUMMARY:
This is a study to collect and bank tissue specimens and blood from patients with Hepatoblastoma.

DETAILED DESCRIPTION:
COG 9346 - Lay Summary

Hepatoblastoma Biology Study and Tissue Bank

Although tremendous improvement in the treatment of childhood cancer has resulted from the use of clinical trials, it is clear that additional significant progress will require a better understanding of the molecular makeup of pediatric malignancies. Hepatoblastoma, an embryonal tumor of the liver, is rare in the general population. It occurs in approximately 1 in 50,000 children. However, families affected with Familial Adenomatous Polyposis, in which there is a high incidence of colon cancer, have an 850 fold increase in the frequency of Hepatoblastoma. Hepatoblastoma also occurs in association with Beckwith-Wiedemann Syndrome. Thus the occurrence of Hepatoblastoma suggests the need for both careful investigations into the family history of malignancies in relatives, as well as a search for genetic alterations that may contribute to tumor development.

COG cancer researchers are trying to better understand the causes of Hepatoblastoma. They want to develop improved methods for treatment, diagnosis and possibly even prevention. The exact molecules or genes to be studied will change over time as progress in cancer research is made. Not every gene or molecule known to be involved in cancer will be studied. Researchers will choose to study only those genes or molecules which they think are most promising. At present, the study of at least three genes is planned.

In some cases these changes may be detected in normal tissues such as liver or blood cells. One of the genes to be studied is known as the APC gene. It is linked with colon cancer in adults. Rarely this gene can be passed on in families which are prone to develop both colon cancer and Hepatoblastoma. We don't know how common changes in this gene are in children with Hepatoblastoma. This study will try and figure out if this gene is commonly changed in Hepatoblastoma.

In addition to studying specific genes or molecules, geneticists (doctors who specialize in looking at genes) will look at the overall genetic content of tumors from some of the children involved in this study. This will be done by what is known as a karyotype or chromosome analysis. It is known that some Hepatoblasomas have extra copies of certain chromosomes. However, we do not know what effect these extra chromosomes might have on predicting which children will be most likely to respond to treatment. One of the goals of the study is to figure out what biological factors within the tumors, including extra chromosomes, might help predict which children will respond best to treatment. This will hopefully lead to better treatment of Hepatoblastoma.

A single extra blood sample will be taken from the patient for this study. We will take no more than 1 1/2 teaspoons of blood. This amount may be less for very small infants. We will also take a single blood sample (1 tablespoon) from the parent.

A portion of tumor tissue that is removed from the patient's surgery or biopsy will also be sent. No extra procedures will be done to get the tumor tissue. It will be taken during a surgery that is needed for standard care.

Patients will also be asked to complete a questionnaire about their background. They may also be asked to complete a follow-up questionnaire or to provide additional information in the future.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hepatoblastoma.

Exclusion Criteria:

-

Ages: 6 Months to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2005-09; Primary Completion 2015-01 (Estimated); Study Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
To collect and bank Hepatoblastoma specimens. | specimens will be banked indefinitely

CONTACTS AND LOCATIONS:
Overall Officials: Howard Katzenstein, MD, Principal Investigator — Children's Healthcare of Atlanta
Locations (1):
- Children's Healthcare of Atlanta, Atlanta, Georgia, United States